CLINICAL TRIAL: NCT03420404
Title: A Pragmatic Randomized Controlled Trial of a Novel TCM Physician-involved Collaborative Care Model in the Management of Patients With Axial Spondyloarthritis in Singapore (AcuSpA)
Brief Title: Clinical Trial of TCM Collaborative Care Model in Axial Spondyloarthritis
Acronym: AcuSpA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Saw Swee Hock School of Public Health (Unknown); National University of Singapore (Other); Thong Chai Medical Institute Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/2088
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The rheumatologist will be blinded for the first 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative care with TCM physicians (Experimental): TCM physician involved collaborative care model (TCMCMC): The intervention arm will involve the TCM physician in the management of patients with AxSpA in addition to the usual rheumatological care.
  Interventions: Other: TCM physician involved collaborative care model (TCMCMC)
- Usual care only (No Intervention): The attending rheumatologist will prescribe a variety of treatment inclusive of medications such as non-steroidal anti-inflammatory drugs and physiotherapy.

INTERVENTIONS:
Other: TCM physician involved collaborative care model (TCMCMC) — TCM physician delivered acupuncture as well as history taking, physical examination, non-pharmacological advice and communications with rheumatologists.
  Acupuncture procedures: After eliciting the deqi sensation, the needles will be left in place for 30 minutes. The acupuncture treatment will be done 2-3 times a week, with 5 sessions constituting a treatment course. There will be a break of 1 week in between each acupuncture course. Patients in the intervention arm will undergo 2 treatment courses (or 10 sessions) in total.
  Arms: Collaborative care with TCM physicians

SUMMARY:
A pragmatic, prospective, randomized controlled trial will be conducted in patients with axial spondyloarthritis who are NSAID inadequate responders. Patients will be randomized in a 1:1 ratio to either receive standard rheumatological care or a Traditional Chinese Medicine physician involved collaborative model of care (i.e. NSAIDs with acupuncture). Primary end-point was spinal pain score at week 6 with secondary end-points being evaluated week 24. Through this study, we hope to assess a novel model of care in AxSpA and be used as a reference to improve the management of other chronic diseases in Singapore.

DETAILED DESCRIPTION:
The objective of this study is to determine the clinical effectiveness, safety and cost-effectiveness of a new model of care in the management of Spondyloarthritis (AxSpA) using a pragmatic trial approach. In this study, we define TCM physician involved collaborative model of care (TCMCMC) as TCM physician delivered acupuncture as well as TCM physician's history taking, physical examination, non-pharmacological advice and communications with rheumatologists in addition to the usual rheumatological care. The TCMCMC involves TCM physicians diagnosing patients based on TCM clinical syndromes and prescribing standardised acupuncture treatment. The patient population will still receive their standard of care (drug therapy and physiotherapy) as background therapy. The proposed study will not be investigating any therapeutic or medicinal products (drugs).

Our primary hypothesis is that novel TCMCMC in patients with AxSpA will result in better pain control as compared the usual rheumatological care. Secondary hypothesis is that TCMCMC will have greater improvements in other clinical, quality of life, and economic outcomes as compared with those under the usual rheumatological care.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Have AxSpA, diagnosed according to the 2009 Assessment of Spondyloarthritis International Society (ASAS) criteria
* Have active disease based on Bath AS Disease Activity Index (BASDAI) score ≥4 on a 11-point Numerical Rating Scale (NRS) and spinal pain score ≥4 on a 11-point NRS
* Has failed 2 sequential NSAIDs (including COX-2 inhibitor) at maximal tolerated doses for ≥ 4 weeks
* No biologic therapy (i.e tumour necrosis factor blocker or anti-interleukin 17) within the past three months
* Patient who is on current treatment with concomitant methotrexate (MTX) or sulfasalazine (SSZ) at study entry must be on the drug for ≥12 weeks and at stable dose for ≥4 weeks prior to randomisation. Patients who are on non-biologic disease-modifying antirheumatic drugs (DMARDs) other than methotrexate or sulfasalazine must discontinue the DMARD 4 weeks prior to randomisation, except for leflunomide, which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine washout has been performed. Patients taking systemic corticosteroids have to be on stable dose of ≤ 10mg/day prednisolone or equivalent for at least two weeks before randomisation

Exclusion Criteria:

* Pregnant or breastfeeding women
* On anti-platelet agents (i.e. aspirin, clopidogrel, dipyridamole, etc) and anti-coagulants (i.e. warfarin, enoxaparin, rivaroxaban, dabigatran, etc)
* Have bleeding disorders
* Have blood-borne communicable diseases (e.g. hepatitis B, hepatitis C, human immunodeficiency virus, etc).

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean difference in spinal pain score | Baseline, Week 6
  Mean difference in spinal pain score between intervention and control groups at week 6 of treatment.

SECONDARY OUTCOMES:
Mean difference in spinal pain score | Baseline, Week 12, Week 24
  Mean difference in spinal pain score between intervention and control groups at week 12 and week 24 of treatment.
Mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline, Week 6, Week 12, Week 24
  Mean difference in BASDAI score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline, Week 6, Week 12, Week 24
  Mean difference in BASFI score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in Bath Ankylosing Spondylitis Global score (BAS-G) | Baseline, Week 6, Week 12, Week 24
  Mean difference in BAS-G score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in Health Assessment Questionnaire (HAQ) | Baseline, Week 6, Week 12, Week 24
  Mean difference in HAQ score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in 36-Item Short Form Survey (SF-36) | Baseline, Week 6, Week 12, Week 24
  Mean difference in SF-36 score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in Ankylosing Spondylitis Quality of Life (ASQoL) | Baseline, Week 6, Week 12, Week 24
  Mean difference in AsQoL score between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in consultation fees (rheumatologist and other outpatient) and drugs | Week 6, Week 12, Week 24
  Mean difference in consultation fees and drugs between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in costs of laboratory procedures and imaging | Week 6, Week 12, Week 24
  Mean difference in costs of laboratory procedures and imaging between intervention and control groups at week 6, week 12 and week 24 of treatment.
Mean difference in number of inpatient days | Week 6, Week 12, Week 24
  Mean difference in number of inpatient days between intervention and control groups at week 6, week 12, week 24 of treatment.

OTHER OUTCOMES:
Mean difference in spinal pain score | Baseline, Week 52
  Mean difference in spinal pain score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline, Week 52
  Mean difference in BASDAI score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline, Week 52
  Mean difference in BASFI score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in Bath Ankylosing Spondylitis Global score (BAS-G) | Baseline, Week 52
  Mean difference in BAS-G score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in Health Assessment Questionnaire (HAQ) | Baseline, Week 52
  Mean difference in HAQ score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in 36-Item Short Form Survey (SF-36) | Baseline, Week 52
  Mean difference in SF-36 score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in Ankylosing Spondylitis Quality of Life (ASQoL) | Baseline, Week 52
  Mean difference in AsQoL score between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in consultation fees (rheumatologist and other outpatient) and drugs | Week 52
  Mean difference in consultation fees and drugs between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in number of inpatient days | Week 52
  Mean difference in number of inpatient days between intervention and control groups at week 52 of treatment will serve as exploratory outcome.
Mean difference in costs of laboratory procedures and imaging | Week 52
  Mean difference in costs of laboratory procedures and imaging between intervention and control groups at week 52 of treatment will serve as exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Fong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meng CF, Wang D, Ngeow J, Lao L, Peterson M, Paget S. Acupuncture for chronic low back pain in older patients: a randomized, controlled trial. Rheumatology (Oxford). 2003 Dec;42(12):1508-17. doi: 10.1093/rheumatology/keg405. Epub 2003 Jul 30. PMID 12890859
- [Derived] Kwan YH, Fong W, Ang XL, Chew XY, Yoon S, Tan CS, Tai BC, Huang Y, Bilger M, Phang JK, Tan HC, Quek SA, Eng SYC, Tan CT, Dong BQ, Koh HL, Leung YY, Ng SC, Fong KY, Thumboo J, Ostbye T. Facilitators of and barriers to implementing a traditional Chinese medicine collaborative model of care for axial spondyloarthritis: a qualitative study. Acupunct Med. 2021 Dec;39(6):629-636. doi: 10.1177/09645284211009543. Epub 2021 May 28. PMID 34049443
- [Derived] Kwan YH, Fong W, Ang XL, Tan CS, Tai BC, Huang Y, Bilger M, Phang JK, Tan HC, Lee JV, Sun L, Tan CT, Dong BQ, Koh HL, Leung YY, Lui NL, Yeo SI, Ng SC, Fong KY, Thumboo J, Ostbye T. Traditional Chinese medicine (TCM) collaborative care for patients with axial spondyloarthritis (AcuSpA): protocol for a pragmatic randomized controlled trial. Trials. 2019 Jan 14;20(1):46. doi: 10.1186/s13063-018-3117-2. PMID 30642381

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03420404/Prot_SAP_003.pdf